CLINICAL TRIAL: NCT07311018
Title: The Effects of Neuromuscular Electrical Stimulation and Leap Motion-Based Exercises on Hand Function Parameters in Cerebral Palsy
Brief Title: Neuromuscular Electrical Stimulation and Leap Motion-Based Exercises in Cerebral Palsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande Özlü Erdoğan, PhD Candidate- MSc. Physiotherapist- Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-3234
Record Dates: First submitted 2025-11-25; First posted 2025-12-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: cerebral palsy; leap motion controller; neuromuscular electrical stimulation; hand function; physiotherapy; virtual reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leap Motion Group (Experimental): Participants in this group will perform upper extremity exercises using the Leap Motion Controller combined with virtual reality-based training, in addition to conventional rehabilitation.
  Interventions: Device: Leap Motion-Based Exercise Program; Behavioral: Conventional Exercise Program
- NMES Group (Experimental): Participants in this group will receive Neuromuscular Electrical Stimulation (NMES) applied to the wrist extensor muscles, in addition to conventional rehabilitation.
  Interventions: Device: NMES; Behavioral: Conventional Exercise Program

INTERVENTIONS:
Device: Leap Motion-Based Exercise Program — Participants assigned to the Leap Motion group will receive Leap Motion-based upper extremity exercise training. The program consists of interactive virtual reality tasks targeting wrist and hand movements. Each session includes 20 minutes of Leap Motion-based exercises, delivered three times per week for 8 weeks. In addition, participants will receive 40 minutes of conventional upper extremity exercises per session (one session is total 60 minutes).
  Arms: Leap Motion Group
Device: NMES — Participants assigned to the NMES group will receive neuromuscular electrical stimulation applied to the wrist extensor muscles. NMES will be administered for 20 minutes per session, three times per week, for 8 weeks, following standard pediatric rehabilitation parameters. Each session will also include 40 minutes of conventional upper extremity exercises ( one session is total 60 minutes).
  Arms: NMES Group
Behavioral: Conventional Exercise Program — All participants will receive routine conventional upper extremity exercises. During the pre-intervention phase, participants will complete a 4-week program consisting of 40 minutes per session, three times per week. During the 8-week intervention period, both groups will continue to receive 40 minutes of conventional exercises in each session.

SUMMARY:
Cerebral palsy (CP) is a group of disorders resulting from a permanent but non-progressive lesion in the developing brain, which affects the development of movement and posture and may lead to activity limitations. Upper extremity involvement is observed in approximately 60% of children with CP. Abnormal muscle tone, imbalance between agonist and antagonist muscles, spasticity, alignment problems, reduced muscle strength, and impaired motor control are among the upper extremity impairments seen in CP. As a result, hand use is typically affected in a way that negatively influences the performance of daily living activities. Upper extremity functionality and hand use are crucial for participation in daily life and overall quality of life in children with CP.

In addition to conventional rehabilitation methods, advances in technology have introduced various new modalities for upper extremity rehabilitation. The aim of the present project is to investigate the effects of Leap Motion-based exercise intervention and Neuromuscular Electrical Stimulation (NMES) on hand functions in children with spastic CP.

A total of 30 children aged 6-15 years with a diagnosis of spastic CP and distal upper extremity involvement will be included in the study. To evaluate eligibility according to the inclusion criteria, gross motor function level will be assessed using the Gross Motor Function Classification System (GMFCS); hand skills will be assessed using the Manual Ability Classification System (MACS); upper extremity muscle tone will be assessed using the Modified Ashworth Scale (MAS); and passive wrist extension range of motion (ROM) will be measured using an electronic goniometer.

Following eligibility confirmation, baseline assessments will be conducted. At baseline wrist ROM will be measured using an electronic goniometer; selective motor control of the wrist will be assessed using the Selective Control of the Upper Extremity Scale (SCUES); hand functions will be evaluated using the Jebsen-Taylor Hand Function Test; daily hand use will be assessed using the ABILHAND-Kids; and wrist extensor and flexor strength and activation will be evaluated via surface electromyography (sEMG).

All participants will then undergo a 4-week routine conventional exercise program (3 sessions per week, 40 minutes per session). At the end of this 4-week period assessments will be repeated (at week 4). Subsequently, the 30 children with CP will be randomly allocated into two groups: the Leap Motion Control group (n = 15) and the NMES group (n = 15). Both groups will receive an 8-week intervention consisting of 3 sessions per week, each lasting 60 minutes (20 minutes of Leap Motion-based exercises or 20 minutes of NMES application, in addition to 40 minutes of conventional exercises). At the end of the 8-week intervention, all assessments will be repeated ( at week 12).

For statistical analyses, the Statistical Package for the Social Sciences (SPSS) Version 23.0 for Windows will be used.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic unilateral or bilateral cerebral palsy based on clinical and MRI findings.
* Involvement of the distal upper extremity (wrist and/or fingers).
* Aged between 6 and 15 years.
* No history of botulinum toxin injection or surgical intervention to the upper extremity within the past 6 months.
* Gross Motor Function Classification System (GMFCS) levels I-III.
* Manual Ability Classification System (MACS) levels I-III.
* Upper extremity spasticity corresponding to 0, 1, or 1+ on the Modified Ashworth Scale (MAS).
* Passive wrist extension limitation not exceeding 10 degrees.
* Ability to follow verbal instructions (mental level reported as "normal" or "mild mental retardation" in the medical record).

Exclusion Criteria:

* Currently participating in a specific hand rehabilitation program.
* Presence of visual or hearing impairment.
* History of epilepsy.
* Presence of chronic, orthopedic, or systemic conditions that may interfere with participation.
* GMFCS levels IV or V.
* MACS levels IV or V.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Hand Function | Baseline (at week 0), after completion of a 4-week conventional exercise program (at week 4), and after completion of an additional 8-week intervention period (at week 12).
  Hand Function will be assessed with Jebsen-Taylor Hand Function Test. JTHFT is a timed, seven-subtest assessment designed to evaluate hand functionality. The test is derived from common daily activities and includes the following tasks: writing a standardized 24-letter sentence, turning five cards, picking up small objects, picking up five beans using a spoon, stacking four checkers on a test board, moving five large empty cans, and moving five full cans. Since the study population includes children who may not yet be literate according to the age criteria, the first subtest (writing a sentence) will be omitted from the evaluation. Each subtest allows a maximum of 120 seconds for successful completion. All subtests are first performed with the non-dominant hand, followed by the dominant hand. For each subtests shorter times indicate better performance. The validity and reliability of the JTHFT in children with cerebral palsy aged 6-18 years have been established by Tofani et al.

SECONDARY OUTCOMES:
Goniometric Assessment | Baseline (at Week 0), after completion of a 4-week conventional exercise program (at Week 4), and after completion of an additional 8-week intervention period (at Week 12).
  Active wrist range of motion (ROM) will be assessed using an electronic goniometer (Baseline Digital Absolute+ Axis), in addition to the Becure HandROM application integrated into the Leap Motion Controller (LMC). Wrist flexion, extension, ulnar deviation, and radial deviation ROM will be measured bilaterally. Each measurement will be repeated three times, and the mean value will be used for statistical analysis.
Selective Motor Control | Baseline (at week 0), after completion of a 4-week conventional exercise program (at week 4), and after completion of an additional 8-week intervention period (at week 12).
  Selective motor control will be assessed with Selective Control of the Upper Extremity Scale (SCUES). SCUES was developed to assess selective voluntary motor control (SVMC) of the upper extremity and represents the first scale specifically designed for this purpose. It is a practical and user-friendly, video-based assessment tool that can be administered in less than 15 minutes. The test provides the opportunity to assess selective movements in all upper extremity joints, including the shoulder, elbow, forearm, wrist, and fingers. Each of the five joint regions is scored on a four-point ordinal scale: absence of SVMC (0 points), moderately reduced SVMC (1 point), mildly reduced SVMC (2 points), and normal SVMC (3 points). The total SCUES score ranges from 0 to 15, with higher scores indicating better SVMC. In the present study, only the selective control of the wrist joint will be assessed bilaterally.
Muscle Activation | Baseline (at week 0), after completion of a 4-week conventional exercise program (at week 4), and after completion of an additional 8-week intervention period (at week 12).
  Surface electromyography (sEMG) is based on the principle that there is a linear relationship between sEMG signal amplitude and muscle contraction force, with signal amplitude increasing as muscle force increases. In the present study, muscle activation will be assessed using the Natus UltraPro® S100 (EMG/NCS/EP neurodiagnostic system). Surface electrodes will be applied to measure muscle activity. The child will be asked to perform maximum voluntary contraction (MVC), and the motor action potentials of the muscles will be recorded for 10-15 seconds, followed by a 10-second rest period. Each measurement will be repeated three times, and activation of the wrist extensor and flexor muscles will be recorded. sEMG assessments will be conducted with the support of neurology specialist.
Hand Use in Daily Activities | Baseline (at week 0), after completion of a 4-week conventional exercise program (at week 4), and after completion of an additional 8-week intervention period (at week 12).
  The ABILHAND-Kids questionnaire will be used to assess hand use in daily life activities. ABILHAND-Kids is designed to measure upper extremity function in children with cerebral palsy aged 6-15 years and to evaluate unimanual and bimanual activities of the upper limbs as comprehensively as possible. The questionnaire consists of 21 items covering both unimanual and bimanual tasks and is completed by the child's parents using a three-point scale: 0-cannot perform the activity, 1-performs the activity with difficulty, and 2-performs the activity easily. Raw scores are converted to Rasch-based logit scores, with higher scores indicating better manual ability. ABILHAND-Kids is a test specifically developed for children with cerebral palsy and requires no preparatory phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Physiotherapy and Rehabilitation Department, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ou CH, Shiue CC, Kuan YC, Liou TH, Chen HC, Kuo TJ. Neuromuscular Electrical Stimulation of Upper Limbs in Patients With Cerebral Palsy: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Am J Phys Med Rehabil. 2023 Feb 1;102(2):151-158. doi: 10.1097/PHM.0000000000002058. Epub 2022 Jun 9. PMID 35687763
- [Background] Rathinam C, Mohan V, Peirson J, Skinner J, Nethaji KS, Kuhn I. Effectiveness of virtual reality in the treatment of hand function in children with cerebral palsy: A systematic review. J Hand Ther. 2019 Oct-Dec;32(4):426-434.e1. doi: 10.1016/j.jht.2018.01.006. Epub 2018 Jul 14. PMID 30017414
- [Background] Schmidt, B. G., Gerzson, L. R., ve Almeida, C. S. D. 2020. "The use of surface electromiography as a measure of physiotherapy outcomes in children with Cerebral Palsy: a systematic review", Journal of Human Growth and Development, 30(2), 216-226.
- [Background] Yildizgoren MT, Nakipoglu Yuzer GF, Ekiz T, Ozgirgin N. Effects of neuromuscular electrical stimulation on the wrist and finger flexor spasticity and hand functions in cerebral palsy. Pediatr Neurol. 2014 Sep;51(3):360-4. doi: 10.1016/j.pediatrneurol.2014.05.009. Epub 2014 May 21. PMID 25011433
- [Background] Tarakci E, Arman N, Tarakci D, Kasapcopur O. Leap Motion Controller-based training for upper extremity rehabilitation in children and adolescents with physical disabilities: A randomized controlled trial. J Hand Ther. 2020 Apr-Jun;33(2):220-228.e1. doi: 10.1016/j.jht.2019.03.012. Epub 2019 Apr 19. PMID 31010703
- [Background] Xu K, He L, Mai J, Yan X, Chen Y. Muscle Recruitment and Coordination following Constraint-Induced Movement Therapy with Electrical Stimulation on Children with Hemiplegic Cerebral Palsy: A Randomized Controlled Trial. PLoS One. 2015 Oct 9;10(10):e0138608. doi: 10.1371/journal.pone.0138608. eCollection 2015. PMID 26452230
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Komariah M, Amirah S, Abdurrahman MF, Handimulya MFS, Platini H, Maulana S, Nugrahani AD, Mulyana AM, Qadous SG, Mediani HS, Mago A. Effectivity of Virtual Reality to Improve Balance, Motor Function, Activities of Daily Living, and Upper Limb Function in Children with Cerebral Palsy: A Systematic Review and Meta-Analysis. Ther Clin Risk Manag. 2024 Feb 14;20:95-109. doi: 10.2147/TCRM.S432249. eCollection 2024. PMID 38375076
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] Herrero P, Carrera P, Garcia E, Gomez-Trullen EM, Olivan-Blazquez B. Reliability of goniometric measurements in children with cerebral palsy: a comparative analysis of universal goniometer and electronic inclinometer. A pilot study. BMC Musculoskelet Disord. 2011 Jul 10;12:155. doi: 10.1186/1471-2474-12-155. PMID 21740600
- [Background] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Background] Cortes-Perez I, Zagalaz-Anula N, Montoro-Cardenas D, Lomas-Vega R, Obrero-Gaitan E, Osuna-Perez MC. Leap Motion Controller Video Game-Based Therapy for Upper Extremity Motor Recovery in Patients with Central Nervous System Diseases. A Systematic Review with Meta-Analysis. Sensors (Basel). 2021 Mar 15;21(6):2065. doi: 10.3390/s21062065. PMID 33804247
- [Background] Surveillance of Cerebral Palsy in Europe. Surveillance of cerebral palsy in Europe: a collaboration of cerebral palsy surveys and registers. Surveillance of Cerebral Palsy in Europe (SCPE). Dev Med Child Neurol. 2000 Dec;42(12):816-24. doi: 10.1017/s0012162200001511. PMID 11132255
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Arnould C, Penta M, Renders A, Thonnard JL. ABILHAND-Kids: a measure of manual ability in children with cerebral palsy. Neurology. 2004 Sep 28;63(6):1045-52. doi: 10.1212/01.wnl.0000138423.77640.37. PMID 15452296
- [Background] Akpinar P, Tezel CG, Eliasson AC, Icagasioglu A. Reliability and cross-cultural validation of the Turkish version of Manual Ability Classification System (MACS) for children with cerebral palsy. Disabil Rehabil. 2010;32(23):1910-6. doi: 10.3109/09638281003763796. PMID 20373857
- [Background] Avcil E, Tarakci D, Arman N, Tarakci E. Upper extremity rehabilitation using video games in cerebral palsy: a randomized clinical trial. Acta Neurol Belg. 2021 Aug;121(4):1053-1060. doi: 10.1007/s13760-020-01400-8. Epub 2020 Jun 11. PMID 32524538
- [Background] Daliri M, Moradi A, Fatorehchy S, Bakhshi E, Moradi E, Sabbaghi S. Investigating the Effect of Leap Motion on Upper Extremity Rehabilitation in Children with Cerebral Palsy: A Randomized Controlled Trial. Dev Neurorehabil. 2023 May;26(4):244-252. doi: 10.1080/17518423.2023.2203210. Epub 2023 Apr 25. PMID 37122098
- [Background] Acikbas, E., Tarakci, D., ve Budak, M. 2020. "Comparison of the effects of Kinesio tape and neuromuscular electrical stimulation on hand extensors in children with cerebral palsy", Int J Ther Rehabil,27:1-12,